CLINICAL TRIAL: NCT04478084
Title: Immunogenicity and Safety of a Purified Vero Rabies Vaccine-Serum Free (VRVg) Assessed With the Institut Pasteur du Cambodge (IPC: 2-2-2-0-0) and the Thai Red Cross (TRC: 2-2-2-0-2) Intradermal Regimens as Simulated Rabies Post-exposure Prophylaxis in Healthy Subjects in Thailand
Brief Title: Study of Purified Vero Rabies Vaccine Compared With a Reference Rabies Vaccine as Simulated Rabies Post-Exposure Prophylaxis in Adult and Pediatric Population in Thaïland
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: VRV09; U1111-1227-4143 (Registry Identifier: ICTRP)
Record Dates: First submitted 2020-07-15; First posted 2020-07-20 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Rabies (Healthy Volunteers)
Keywords: Rabies Vaccine
MeSH Terms: conditions — Rabies

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Modified double-blind: the participant (or legally acceptable representative) and the Investigator remain unaware of the treatment assignments throughout the study. An unblinded qualified trial staff member will prepare and administer the appropriate vaccine but will not be involved in the immunogenicity and safety evaluations.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Group 1: pediatric participants; VRVg-2 (Experimental): VRVg-2 8 injections: 2 at Day 0, 2 at Day 3, 2 at Day 7, and 2 at Day 28
  Interventions: Biological: Purified vero rabies vaccine - serum free VRVg-2
- Group 2: pediatric participants; Verorab (Active Comparator): Verorab 8 injections: 2 at Day 0, 2 at Day 3, 2 at Day 7, and 2 at Day 28
  Interventions: Biological: Purified inactivated rabies vaccine
- Group 3: adult participants; VRVG-2 + ERIG (Experimental): VRVg-2 8 injections: 2 at Day 0, 2 at Day 3 and 2 at Day 7
  + ERIG at D0
  Interventions: Biological: Purified vero rabies vaccine - serum free VRVg-2; Biological: Equine rabies immunoglobulins (ERIG) (only Group 3 and Group 4)
- Group 4: adult participants; Verorab + ERIG (Active Comparator): Verorab 8 injections: 2 at Day 0, 2 at Day 3 and 2 at Day 7
  + ERIG at D0
  Interventions: Biological: Purified inactivated rabies vaccine; Biological: Equine rabies immunoglobulins (ERIG) (only Group 3 and Group 4)
- Group 5: adult participants; VRVG-2 + HRIG (Experimental): VRVg-2 8 injections: 2 at Day 0, 2 at Day 3, 2 at Day 7, and 2 at Day 28
  + HRIG at D0
  Interventions: Biological: Purified vero rabies vaccine - serum free VRVg-2; Biological: Human rabies immunoglobulins (HRIG) (only Group 5 and Group 6)
- Group 6: adult participants; Verorab + HRIG (Active Comparator): Verorab 8 injections: 2 at Day 0, 2 at Day 3, 2 at Day 7, and 2 at Day 28
  + HRIG at D0
  Interventions: Biological: Purified inactivated rabies vaccine; Biological: Human rabies immunoglobulins (HRIG) (only Group 5 and Group 6)

INTERVENTIONS:
Biological: Purified vero rabies vaccine - serum free VRVg-2 — Pharmaceutical form:freeze-dried Route of administration: intradermal
  Arms: Group 1: pediatric participants; VRVg-2; Group 3: adult participants; VRVG-2 + ERIG; Group 5: adult participants; VRVG-2 + HRIG
Biological: Purified inactivated rabies vaccine — Pharmaceutical form:freeze-dried Route of administration: intradermal
  Other Names: Verorab®
  Arms: Group 2: pediatric participants; Verorab; Group 4: adult participants; Verorab + ERIG; Group 6: adult participants; Verorab + HRIG
Biological: Equine rabies immunoglobulins (ERIG) (only Group 3 and Group 4) — Pharmaceutical form: liquid/solution in 5 mL vials Route of administration: intramuscular
  Other Names: ERIG
  Arms: Group 3: adult participants; VRVG-2 + ERIG; Group 4: adult participants; Verorab + ERIG
Biological: Human rabies immunoglobulins (HRIG) (only Group 5 and Group 6) — Pharmaceutical form: liquid/solution in 2 mL vials Route of administration: intramuscular
  Other Names: IMOGAM® Rabies-HT
  Arms: Group 5: adult participants; VRVG-2 + HRIG; Group 6: adult participants; Verorab + HRIG

SUMMARY:
Primary Objective:

To describe the immune response induced by VRVg-2 and Verorab vaccine at Day 14 (to assess the immune response after 3 doses [2-2-2]) and Day 42 (to assess the immune response after 4 doses [2-2-2-0-2]) when administered as standalone in healthy pediatric population or co-administered with HRIG (Group 5 and Group 6) at Day 0 in healthy adults.

Secondary Objectives:

* To describe the immune response induced by VRVg-2 and Verorab vaccine at Day 14 (to assess the immune response after 3 doses [2-2-2]) when co-administered with ERIG (Group 3 and Group 4) at Day 0 in healthy adults
* To describe the immune response induced by VRVg-2 and Verorab vaccine at D90 (to assess the immune response 90 days post-rabies simulated exposure) when administered as standalone in healthy pediatric population or co-administered with HRIG (Group 5 and Group 6) at Day 0 in healthy adults
* To describe the safety profile of VRVg-2 and Verorab vaccine as standalone in pediatric population or when co-administered with ERIG (Group 3 and Group 4) or HRIG (Group 5 and Group 6) at Day 0 in adults, after each vaccination.

DETAILED DESCRIPTION:
The duration of each participant's participation in the study is approximately 7 months (28 day-vaccination period followed by 6 month safety follow-up period).

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria :

* Aged ≥ 1 year on the day of inclusion
* Participant (adult ≥ 18 years without upper age limit) or participant and participant's parent/LAR (child ≥ 1 to < 18 years) are able to attend all scheduled visits and to comply with all study procedures

The following criterion only applies to healthy adults ≥ 18 years:

- Body Mass Index (BMI): 18.5 kg/m2 ≤ BMI ≤ 30 kg/m2

Exclusion Criteria:

Exclusion criteria:

* Pregnant, or lactating, or of childbearing potential and not using an effective method of contraception or abstinence from at least 4 weeks prior to the first vaccination and until 1 month after each vaccination. To be considered of non-childbearing potential, a female must be pre-menarche or post-menopausal for at least 1 year, or surgically sterile.
* Participation at the time of study enrollment or, planned participation during the present study period in another clinical study investigating a vaccine, drug, medical device, or medical procedure
* Receipt of any vaccine in the 4 weeks (28 days) preceding the first study vaccination or planned receipt of any vaccine prior to Visit 8 (D90)
* Previous vaccination against rabies (in pre- or post-exposure regimen) with either the study vaccines or another vaccine
* Bite by, or exposure to a potentially rabid animal in the previous 6 months without post-exposure prophylaxis
* Receipt of immune globulins, blood or blood-derived products in the past 3 months
* Known or suspected congenital or acquired immunodeficiency; or receipt of immunosuppressive therapy, such as anti-cancer chemotherapy or radiation therapy, within the preceding 6 months; or long-term systemic corticosteroid therapy (prednisone or equivalent for more than 2 consecutive weeks within the past 3 months)
* At high risk for rabies exposure
* Known systemic hypersensitivity to any of the study/control vaccine components or, for adults, to ERIG Group 3 and Group 4) or HRIG (Group 5 and Group 6), or history of a life-threatening reaction to the vaccines used in the study or to a vaccine containing any of the same substances
* Positive skin test to ERIG at Visit 1 for only adult participants enrolled in Group 3 and Group 4 as per superseded Protocol version 5.0
* Self-reported thrombocytopenia
* Bleeding disorder, or receipt of anticoagulants in the 3 weeks preceding inclusion
* Deprived of freedom by an administrative or court order, or in an emergency setting, or hospitalized involuntarily
* Current alcohol or substance abuse that, in the opinion of the Investigator, might interfere with the study conduct or completion
* Chronic illness that, in the opinion of the Investigator, is at a stage where it might interfere with study conduct or completion
* Moderate or severe acute illness/infection (according to Investigator judgment) on the day of vaccination or febrile illness (temperature ≥ 38.0 C). A prospective subject should not be included in the study until the condition has resolved or the febrile event has subsided
* Personal history of Guillain-Barré syndrome
* Identified as an Investigator or employee of the Investigator or study center with direct involvement in the proposed study, or identified as an immediate family member (ie, parent, spouse, natural or adopted child) of the Investigator or employee with direct involvement in the proposed study
* Receipt of chloroquine or hydroxychloroquine up to 2 months prior to the study or through to study until Visit 8

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 1 Year | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 403 (Actual)
Dates: Start 2020-08-04 (Actual); Primary Completion 2022-03-19 (Actual); Study Completion 2022-07-21 (Actual)

PRIMARY OUTCOMES:
Percentage of participants in Group 1, Group 2, Group 5 and Group 6 achieving rabies virus neutralizing antibody (RVNA) titer greater than or equal to (≥) 0.5 IU/mL | Day 14 (post-vaccination)
  RVNA titers will be measured by rapid fluorescent focus inhibition test (RFFIT)
Percentage of participants in Group 1, Group 2, Group 5 and Group 6 achieving RVNA titer greater than or equal to (≥) 0.5 IU/mL | Day 42 (post-vaccination)
  RVNA titers will be measured by RFFIT
Number of Participants in Group 1, Group 2, Group 5 and Group 6 achieving RVNA titer greater than or equal to (≥) lower limit of quantification | Day 14 (post-vaccination)
  RVNA titers will be measured by RFFIT Lower limit of quantification for RFFIT assay is 0.2 IU/mL
Number of Participants in Group 1, Group 2, Group 5 and Group 6 achieving RVNA titer greater than or equal to (≥) lower limit of quantification | Day 42 (post-vaccination)
  RVNA titers will be measured by RFFIT Lower limit of quantification for RFFIT assay is 0.2 IU/mL
Geometric Mean Titer Ratio (GMTR) of individual RVNA titer: (post-/pre-vaccination) in Group 1, Group 2, Group 5 and Group 6 Participants | Day 14 (post-vaccination)
  RVNA titers against rabies virus will be measured by RFFIT at Day 0 and Day 14 RVNA ratios Day14/Day0 will be calculated
Geometric Mean Titer Ratio (GMTR) of individual RVNA titer: (post-/pre-vaccination) in Group 1, Group 2, Group 5 and Group 6 Participants | Day 42 (post-vaccination)
  RVNA titers against rabies virus will be measured by RFFIT at Day 0 and Day 42 RVNA ratios Day42/Day0 will be calculated

SECONDARY OUTCOMES:
Number of participants reporting immediate adverse events (AEs) | Within 30 minutes post-vaccination
  Includes unsolicited (spontaneously reported) systemic AEs
Percentage of participants reporting solicited injection site reactions | Within 7 days post-vaccination
  Solicited injection site reactions:
  * tenderness, erythema, swelling in toddlers (aged ≥ 1 year to < 2 years)
  * pain, erythema, and swelling in children (aged 2 years to < 12 years), in adolescents and adults (aged ≥ 12 years)
Percentage of participants reporting solicited systemic reactions | Between Day 0 and Day 3, between Day 3 and Day 7, and during the 7 days following the remaining vaccinations
  Solicited systemic reactions:
  * fever, vomiting, crying abnormal, drowsiness, appetite lost, irritability in toddlers (aged ≥ 1 year to < 2 years)
  * fever, headache, malaise and myalgia in children (aged 2 years to < 12 years), adolescents or adults (aged ≥ 12 years)
Number of participants reporting unsolicited injection site AEs | Within 28 days post-vaccination
  Unsolicited (spontaneously reported) injection site AEs
Number of participants reporting unsolicited systemic AEs | Between each vaccination and up to 28 days after the last vaccination
  Unsolicited (spontaneously reported) systemic AEs
Number of participants reporting serious adverse events (SAEs) | Up to 6 months post-vaccination
  SAEs, including adverse event of special interest (AESIs)
Percentage of participants in Group 3 and Group 4 achieving rabies virus neutralizing antibody (RVNA) titer greater than or equal to (≥) 0.5 IU/mL | Day 14 (post-vaccination)
  RVNA titers will be measured by RFFIT
Number of Participants in Group 3 and Group 4 achieving RVNA titer greater than or equal to (≥) lower limit of quantification | Day 14 (post-vaccination)
  RVNA titers will be measured by RFFIT Lower limit of quantification for RFFIT assay is 0.2 IU/mL
Geometric Mean Titer Ratio (GMTR) of individual RVNA titer: (post-/pre-vaccination) in Group 3 and Group 4 Participants | Day 14 (post-vaccination)
  RVNA titers against rabies virus will be measured by RFFIT at Day 0 and Day 14 RVNA ratios Day14/Day0 will be calculated
Percentage of participants in Group 1, Group 2, Group 5 and Group 6 achieving rabies virus neutralizing antibody (RVNA) titer greater than or equal to (≥) 0.5 IU/mL | Day 90 (post-vaccination)
  RVNA titers will be measured by RFFIT
Number of Participants in Group 1, Group 2, Group 5 and Group 6 achieving RVNA titer greater than or equal to (≥) lower limit of quantification | Day 90 (post-vaccination)
  RVNA titers will be measured by RFFIT Lower limit of quantification for RFFIT assay is 0.2 IU/mL
Geometric Mean Titer Ratio (GMTR) of individual RVNA titer: (post-/pre-vaccination) in Group 1, Group 2, Group 5 and Group 6 Participants | Day 90 (post-vaccination)
  RVNA titers against rabies virus will be measured by RFFIT at Day 0 and Day 90 RVNA ratios Day90/Day0 will be calculated

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi Pasteur, a Sanofi Company
Locations (3):
- Thailand (3):
  - Investigational Site Number :7640004, Bangkok
  - Investigational Site Number :7640002, Bangkok
  - Investigational Site Number :7640003, Khon Kaen

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- See also: VRV09 Plain Language Results Summary — https://www.trialsummaries.com/Study/StudyDetails?id=25382&tenant=MT_SNY_9011